CLINICAL TRIAL: NCT07247617
Title: Semi-rigid Ureteroscopy Versus Flexible Ureteroscopy in Upper Third Ureteric Stones Management: a Prospective Randomized Trial
Brief Title: Flexible vs Semi-rigid URS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Ahmed Hamada Ali, Urology Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Upper third ureteric stones
Record Dates: First submitted 2025-09-22; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Ureteric Stone; Flexible Ureteroscopy; Upper Urinary Tract Stones
MeSH Terms: conditions — Ureterolithiasis; Urinary Calculi

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexible Ureteroscopy (Active Comparator)
  Interventions: Procedure: Flexible URS
- Semi-Rigid Ureteroscopy (Experimental)
  Interventions: Procedure: Semi-Rigid URS

INTERVENTIONS:
Procedure: Flexible URS — Flexible URS
  Arms: Flexible Ureteroscopy
Procedure: Semi-Rigid URS — Semi-Rigid URS
  Arms: Semi-Rigid Ureteroscopy

SUMMARY:
To compare the efficacy, safety, success rate, operative time, and cost-effectiveness of flexible ureteroscopy versus semirigid ureteroscopy in the management of upper ureteric stones smaller than 2 cm.

The investigators' main concern in this study is Upper third ureteric stones to determine which cases can be treated with Semi-Rigid Ureteroscopy, and which one needs flexible ureteroscopy. This depends on several factors:

1. Division of the upper third of the ureter
2. Stone size
3. Stone impaction
4. Surgeon experience
5. Anesthesia
6. Ureteric dilatation above the stone
7. Mini endoscopy

DETAILED DESCRIPTION:
Ureteroscopy (URS) is a widely accepted minimally invasive approach for treating ureteric stones, particularly proximal (upper) ureteral stones. Options include rigid, semirigid (often grouped as one), and flexible ureteroscopes. Flexible ureteroscopy allows deflection and access to the proximal ureter and intrarenal collecting system, facilitating treatment of stones that are difficult to reach with rigid ureteroscopes due to anatomical constraints or stone migration. Semirigid ureteroscopy has shown good efficacy, particularly for stones amenable to direct access without complex deflection, offering shorter operative times and lower costs. Studies report stone-free rates of approximately 90-93% for flexible URS and 81-90% for semirigid URS, with flexible URS having somewhat higher success in accessing stones and managing fragment migration. However, flexible URS typically incurs higher costs and longer operative times. Semirigid ureteroscopy is often the initial approach for upper ureteric stones where anatomy, stone size (<2 cm), and location allow straightforward access.

* Flexible ureteroscopy is preferred when stones are located higher in the ureter, difficult to reach by semirigid scopes, or if stone migration into the kidney occurs. It is also favored when more maneuverability is required to treat complex anatomy or large stones.
* Both modalities use holmium laser lithotripsy for stone fragmentation.
* Treatment choice also depends on surgeon preference, availability of equipment, and cost considerations.

Despite advances, there is ongoing debate about the optimal first-line ureteroscopic approach for upper ureteric stones, balancing efficacy, safety, cost, and procedure time. Comparing flexible and rigid/semirigid ureteroscopy outcomes informs treatment algorithms, improving patient care and resource utilization, especially in differing healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years
* upper ureteric stone
* ≤20 mm

Exclusion Criteria:

* Associated renal stones
* Any contraindications to Anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
- Stone-free rate at 3 months duration | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut Hospital, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Granholm L, Svendgaard N. Hydrocephalus following traumatic head injuries. Scand J Rehabil Med. 1972;4(1):31-4. No abstract available. PMID 4220357